CLINICAL TRIAL: NCT04490746
Title: Identifcation of Biomarkers for Active Pulmonary Tuberculosis Using a Metabolomics Approach: a Prospective Multicenter Study
Brief Title: Identifcation of Biomarkers for Active Pulmonary Tuberculosis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 研2020-556
Record Dates: First submitted 2020-07-26; First posted 2020-07-29 (Actual); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Tuberculosis; Diagnosis
MeSH Terms: conditions — Tuberculosis; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- active: patients with active tuberculosis
  Interventions: Other: with no intervention, Collect samples
- latent: patients with latent tuberculosis infection
  Interventions: Other: with no intervention, Collect samples
- negtive control: healthy volunteers
  Interventions: Other: with no intervention, Collect samples

INTERVENTIONS:
Other: with no intervention, Collect samples — only with observation,there is no need to intervene

SUMMARY:
This experiment is designed to analyze the metabolites in body fluids from patients with active tuberculosis and latent tuberculosis infection also with health volunteer, then combine the metabolic product features with clinical characteristics, to develop a kind of metabolites targets to evaluate the progress in tuberculosis, thus provide a basis for further utilization of humoral metabolites in the diagnosis of tuberculosis.

ELIGIBILITY:
Inclusion Criteria:

* patients with active tuberculosis and latent tuberculosis infection

Exclusion Criteria:

* have other serious health problems

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: patients with active tuberculosis and latent tuberculosis infection
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-10-01 (Estimated); Primary Completion 2022-10-01 (Estimated); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
metabolic product | 24 hours after sampling
  features up-regulated or down-regulated

CONTACTS AND LOCATIONS:
Overall Officials: Pintong Huang, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- Department of Ultrasound, Second Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Yes
individual participant data (IPD) can be shared after the main unit publish articals
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: by request
Access Criteria: by request